CLINICAL TRIAL: NCT03797482
Title: A Prospective Evaluation of the Peri-operative Hypoxia in Breast Cancer
Acronym: Hypoxia
Status: Recruiting | Type: Observational
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Rajendra A. Badwe, Director, Tata Memorial Centre and Professor, Department of Surgical Oncology, Tata Memorial Centre
Other Study IDs: Protocol 254
Record Dates: First submitted 2018-06-28; First posted 2019-01-09 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Breast cancer tumor tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Intra-operative tumour tissue biopsies: Intra-operative tumour tissue biopsies will be collected for all patients
  Interventions: Procedure: Intra-operative Tumor Tissue Biopsy

INTERVENTIONS:
Procedure: Intra-operative Tumor Tissue Biopsy — The changing pattern of gene expression during surgery has never been studied. This could be an effect of acute hypoxia that sets in the tumour during surgery or could be a surgical response. To study these changes happening in the tumour during surgery, we are taking serial biopsies during surgery, one at the beginning, one midway during surgery and one at the end of surgery. These samples will be snap frozen and stored at -80 deg celsius in biorepository for future analysis.
  Other Names: Breast cancer surgery

SUMMARY:
To understand the effects induced by acute hypoxia that sets in during surgery in breast cancer. To study this, clinical samples (Tumor biopsies) will be obtained during the surgery after partial devascularisation (sample B) and stored for future genomic and proteonomic evaluations.

DETAILED DESCRIPTION:
Three tumor samples will be obtained after the patient is under anaesthesia,

1. Prior to starting surgery (Sample A)
2. The middle intra-operative sample, which will be collected when half the tumour has been devascularized (i.e., somewhere midway during the surgery). (Sample B)
3. A third post excision (anoxic sample C). These tumour tissue samples will be stored as snap frozen, in RNA later and as paraffin sections.

To understand the effects induced by acute hypoxia that sets in during surgery in breast cancer. To study this, clinical samples (Tumor biopsies) will be obtained during and stored for future genomic and proteonomic evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosis of breast cancer (by FNAC or Biopsy)
2. Not received any chemotherapy or surgical intervention except core biopsy.
3. Planed for Breast cancer surgery
4. Willing to give consent for the study

Exclusion Criteria:

1. Clinically diagnosis of Metastatic breast cancer
2. Received any anticancer therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women diagnosed with breast cancer, undergoing surgery upfront
Study Population: Women diagnosed with breast cancer at outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-11-27 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Gene expression changes | The study aims to evaluate gene expression changes during surgical resection, which lasts for 30-90 minutes on an average. Thus, we have not planned a clinical follow-up or collection of data for the patients post sampling during surgical resection.
  The primary outcome measured will be gene expression changes during surgical resection. Messenger ribonucleic acid (mRNA) transcripts will be quantitated and their levels evaluated during different time-points of surgical resection, using high throughput omics technologies (Next generation sequencing, nanostring ncounter, qRT-PCR array).

SECONDARY OUTCOMES:
Immunohistochemistry for other markers | The study aims to evaluate gene expression changes during surgical resection, which lasts for 30-90 minutes on an average. Thus, we have not planned a clinical follow-up or collection of data for the patients post sampling during surgical resection.
  The secondary outcome measured will be protein expression changes during surgical resection. Protein levels will be quantitated, and their levels evaluated, during different time-points of surgical resection. Transcripts found to be de-regulated or changed at different time-points of surgical resection will be evaluated using IHC at protein level. We will also use high throughput omics technologies (SILAC, ITRAQ) for characterising these changes at protein levels.

CONTACTS AND LOCATIONS:
Overall Officials: Rajendra Badwe, Principal Investigator — Director, tata Memorial Centre
Locations (1):
- Tata Memorial Center, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Semenza GL. Cancer-stromal cell interactions mediated by hypoxia-inducible factors promote angiogenesis, lymphangiogenesis, and metastasis. Oncogene. 2013 Aug 29;32(35):4057-63. doi: 10.1038/onc.2012.578. Epub 2012 Dec 10. PMID 23222717
- [Background] Hockel M, Vaupel P. Biological consequences of tumor hypoxia. Semin Oncol. 2001 Apr;28(2 Suppl 8):36-41. PMID 11395851
- [Background] Hoesel B, Schmid JA. The complexity of NF-kappaB signaling in inflammation and cancer. Mol Cancer. 2013 Aug 2;12:86. doi: 10.1186/1476-4598-12-86. PMID 23915189